CLINICAL TRIAL: NCT00791934
Title: Clinical Study of Safety and Efficacy for the Relieva Stratus With Elution of Triamcinolone Acetonide (Kenalog-40)
Brief Title: Clinical Study of Safety and Efficacy for the Relieva Stratus With Elution of Triamcinolone Acetonide
Acronym: DELIVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPR005003
Record Dates: First submitted 2008-11-13; First posted 2008-11-17 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stratus Microflow Ethmoid Spacer (Experimental): Temporary implantation of Ethmoid spacer with Triamcinolone Acetonide for 28 days.
  Interventions: Device: Stratus Microflow Ethmoid Spacer

INTERVENTIONS:
Device: Stratus Microflow Ethmoid Spacer — The Spacer is inserted surgically into the ethmoid complex through the use of a sinus access system. Triamcinolone acetonide will be administered into the Spacer for this investigational study. The Spacer will be left in the ethmoid sinus for a period of 28 days. At the end of the implant period, the device is removed with standard instrumentation, during a follow-up office visit.
  Other Names: Ethmoid Spacer

SUMMARY:
Study Design:

A non-randomized, multi-center, prospective, clinical study intended to evaluate the safety and efficacy of treating the ethmoid sinuses with the Ethmoid Sinus Spacer and Access System used for the local delivery of Triamcinolone Acetonide, over a period of 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects age 17 years or older
* Radiographic evidence of ethmoid disease (baseline CT scan obtained within 30 days of scheduled surgery)
* Diagnosis of chronic sinusitis and failed medical management (minimum of 3 weeks of antibiotics)

Exclusion Criteria:

* Age < 17 years old
* History of glaucoma or diagnosis of glaucoma (baseline visual exam indicating IOP >21 mmHg)
* Adequate anatomical distances for treatment
* Patient received oral steroid treatment within two weeks prior to day of surgery
* Radiographic evidence of extensive sinonasal osteoneogenesis which could prevent device placement
* Sinonasal tumors or obstructive lesions
* History of facial trauma that distorts sinus anatomy and precludes access to the ethmoid sinus
* Contracted/underdeveloped ethmoid sinus
* Dehiscent lamina orbitalis
* Previous ethmoid surgery
* Ethmoid mucocele
* Extensive Nasal Polyps
* Asthmatic patients with aspirin sensitivity
* Pregnant or lactating females

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Catalano, MD, Principal Investigator — Lahey Clinic
Locations (1):
- Lahey Clinic, Burlington, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Stratus Microflow Ethmoid Spacer: Stratus Microflow Ethmoid Spacer: Temporary implantation of the Stratus Microflow Ethmoid Spacer in the ethmoid sinuses with triamcinolone acetonide for a period of 28 days.
Period: Overall Study
Arm/Group | Stratus Microflow Ethmoid Spacer
Started | 63
Completed | 48 (Follow-up extended to 1 yr. 13 subjects chose not to participate in the extension.)
Not Completed | 15
Not completed — Withdrawal by Subject | 2
Not completed — Did not consent for extended follow-up | 13

BASELINE CHARACTERISTICS:
Arm/Group | Stratus Microflow Ethmoid Spacer
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.24 (14.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 58
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Mean Intrapatient Change in Ethmoid Lund-MacKay CT Score (Ethmoid Score Only) at 10 Weeks Post-procedure Compared to Baseline.
Description: The Lund-MacKay (LMK) CT (computed tomography) scoring system is used to evaluate radiographic opacification of the paranasal sinuses, an indicator of sinus disease. The LMK scoring system rates each of both the left and right frontal, maxillary, sphenoid, ostiomeatal complex, anterior ethmoid and posterior ethmoid sinuses on a scale of 0 to 2, where '0' is 'no opacification' and '2' is 'complete opacification'. For this study endpoint, only the ethmoid sinus scores will be evaluated and totaled (left and right anterior and posterior ethmoid sinuses) where zero is the minimum score, and 8 is the maximum score. A higher score represents greater sinus disease burden. The LMK score will be evaluated at 10 weeks post-procedure compared to baseline.
Time Frame: 10 weeks post-procedure
Population: A total of 58 of the 63 subjects had paired baseline and 10 week post-procedure CT scans available for analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Stratus Microflow Ethmoid Spacer
Number analyzed (Participants) | 58
scores on a scale | -1.91 (1.94)

2. Secondary Outcome: Number of Participants With Decrease in Vision Greater Than 2 Lines Per Snellen Chart (BCVA at Baseline vs. BCVA 10 Week Post-procedure)
Description: The Snellen eye chart will be used to evaluate participant's best-corrected visual acuity (BCVA, or best distance vision with eyeglasses or contact lenses) at baseline and at 10 week post-procedure. The number of participants with a decrease in vision greater than 2 lines per the Snellen eye chart are reported for this study endpoint.
Time Frame: 10 weeks post surgery
Population: The analysis population includes paired data for 53 subjects with baseline and 10 week visual acuity data available for analysis.
Measure: Number; unit: participants
Arm/Group | Stratus Microflow Ethmoid Spacer
Number analyzed (Participants) | 53
participants | 0

3. Secondary Outcome: Number of Participants With Either a Change in Intraocular Pressure (IOP) ≥10mmHg OR Documented IOP > 21 mmHg
Description: Change in Intra-Ocular Pressure (IOP) of ≥ 10mmHg or documented IOP of > 21 mmHg were considered clinically significant (baseline compared to 10 weeks post-procedure).
Time Frame: 10 weeks post-procedure
Population: The analysis population includes paired data for 53 of the 63 subjects with intraocular pressure (IOP) evaluations available for analysis.
Measure: Number; unit: participants
Arm/Group | Stratus Microflow Ethmoid Spacer
Number analyzed (Participants) | 53
participants | 1

4. Secondary Outcome: Mean Intra-patient Change in SNOT-20 Score Post-procedure Compared to Baseline
Description: The 20 question Sino-Nasal Outcome Test (SNOT-20) will be used to evaluate sinus symptoms and sinus-symptom related quality of life (QOL) at baseline, 10 weeks, and 1 year post-procedure. The change in SNOT-20 score at each post-procedure time point will be evaluated compared to baseline SNOT-20 score. Each of the 20 questions in the SNOT-20 survey is scored on a scale of 0 to 5, where '0' represents 'no problem' and '5' represents 'problem as bad as it can be'. The 20 questions are expressed as a mean of the scores. Therefore, the minimum mean score is zero and the maximum mean score is 5.
Time Frame: 1 year
Population: The analysis population consists of the 47 subjects with 1 year post-procedure SNOT-20 scores.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Stratus Microflow Ethmoid Spacer
Number analyzed (Participants) | 47
scores on a scale | -1.36 (1.27)

5. Secondary Outcome: Mean Intra-patient Change in SNOT-20 Score Post-procedure Compared to Baseline
Description: as for outcome 4
Time Frame: 10 weeks
Population: The analysis population consists of the 58 subjects with 10 week post-procedure SNOT-20 scores available for analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Stratus Microflow Ethmoid Spacer
Number analyzed (Participants) | 58
scores on a scale | -1.54 (0.99)

ADVERSE EVENTS:
Time Frame: Up to 10 weeks
Description: Adverse event assessment by physician according to defined follow-up visit schedule, and by patient self-reporting
Groups:
- Stratus Microflow Ethmoid Spacer: Temporary implantation of the Stratus Microflow Ethmoid Spacer in the ethmoid sinuses with triamcinolone acetonide for a period of 28 days
Arm/Group | Stratus Microflow Ethmoid Spacer
Serious Adverse Events (participants affected / at risk) | 2/63
Other Adverse Events (participants affected / at risk) | 19/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratus Microflow Ethmoid Spacer (N=63)
Wing Detachment from device (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Device wing separated from the body of the device.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratus Microflow Ethmoid Spacer (N=63)
Headache (Nervous system disorders) | 5 (5) — Adverse event assessment by physician according to defined follow-up visit schedule, and by patient self-reporting.
Nasal Pain (Respiratory, thoracic and mediastinal disorders) | 12 (14) — Adverse event assessment by physician according to defined follow-up visit schedule, and by patient self-reporting.
Nasal Stuffiness (Respiratory, thoracic and mediastinal disorders) | 14 (17) — Adverse event assessment by physician according to defined follow-up visit schedule, and by patient self-reporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days